CLINICAL TRIAL: NCT02823912
Title: Effect of Administration of Capsaicin on Inflammatory Cytokines Profile(TNFα , IL - 1β , IL - 6, IL -8 , MIP - 1β) in Individuals With Dyslipidemia.
Brief Title: Capsaicin Effect on Cytokines Profile in Dyslipidemia
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Guadalajara (Other)
Collaborators: PhD. Teresa Arcelia Garcia Cobian (Unknown); LN. Jessica Lucia Barajas Vega (Unknown)
Responsible Party: Principal Investigator, Ernesto Javier Ramirez Lizardo, PhD., University of Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Capdis
Record Dates: First submitted 2016-07-01; First posted 2016-07-06 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Dyslipidemia; Overweight or Obesity
Keywords: Capsaicin; Dyslipidemia; Inflammatory cytokines
MeSH Terms: conditions — Dyslipidemias; Overweight; Obesity | interventions — Capsaicin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Capsaicin (Experimental): 75 mg capsaicin every 12 hours for 90 days
  Interventions: Drug: Capsaicin
- Control (Placebo Comparator): 75 mg magnesia calcinada every 12 hours for 90 days
  Interventions: Drug: Magnesia calcinada

INTERVENTIONS:
Drug: Capsaicin
  Other Names: Capsicum
  Arms: Capsaicin
Drug: Magnesia calcinada
  Arms: Control

SUMMARY:
The increased mortality from cardiovascular disease has a significant impact on the population, and the prevalence of these diseases it become one of the major problems, since it is the leading cause of mortality and 1 in 3 Mexicans suffer from cardiovascular disease according ENSANUT; the above is attributed to the increase of diseases associated with an inflammatory process accelerated as obesity, dyslipidemia, hypertension (SAH) and diabetes mellitus (DM).

The cholesterol is a major risk factor in the development of cardiovascular disease, and in turn increases the chances of death; however, the treatment of choice is based on changes in lifestyle, which for most people are difficult to maintain long-term. As for the drug therapy treated with drugs many people do not achieve their therapeutic goals, and therefore the inflammatory condition that underlies this disease remains.

Recent studies have focused on the possible role of capsaicin in the inflammatory state through the agonistic effect it has on TRPV1. It has demonstrated the antiinflammatory activity of capsaicin to enhance inflammation by free fatty acids (FFA) and reducing the expression of certain genes involved in this process induced. Capsaicin is a natural choice and well tolerated with few side effects limited to the gastrointestinal tract such as dyspepsia and intestinal irregularity, for the above is of interest to evaluate the effect of capsaicin on the profile of inflammatory cytokines in individuals with dyslipidemia.

DETAILED DESCRIPTION:
It will conduct a clinicala trial, double - blind, randomized and placebo control group. Female and male patients, with dyslipidemia. Two groups will be formed with 17 patients each (capsaicin 150 mg per day or Magnesia calcinada). At the beginning and end of the intervention clinical and laboratory determination. The data obteined were analyzed using SPSS statistical software version 22. It was considered statistically significant at p <0.05

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of dyslipidemia at the time of screening
* BMI of 25 kg /m2 to 34.9 kg / m2
* Without drug treatment in the last three months
* Signature of consent information in writing

Exclusion Criteria:

* Pregnant or lactating
* Total cholesterol ≥ 239 mg / dL, ≥400 TG, LDL-C ≥139
* Other inflammatory diseases
* consumption of some type of supplement
* Diagnosis or history of kidney or liver disease ∞ History of hypersensitivity to the compounds used in the study

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-04 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Inflammatory cytokines profile | 90 days
  TNFα
Inflammatory cytokines profile | 90 days
  IL-1β
Inflammatory cytokines profile | 90 days
  IL-6
Inflammatory cytokines profile | 90 days
  IL-8
Inflammatory cytokines profile | 90 days
  MIP-1β

SECONDARY OUTCOMES:
Lipids profile | 90 days
  total cholesterol
Lipids profile | 90 days
  triglycerides
Lipids profile | 90 days
  C-HDL
Lipids profile | 90 days
  C-LDL
Lipids profile | 90 days
  C-VLDL

CONTACTS AND LOCATIONS:
Overall Officials: Ernesto J Ramirez Lizardo, PhD, Principal Investigator — University Guadalajara

IPD SHARING:
Plan to Share IPD: No